CLINICAL TRIAL: NCT06598748
Title: Effect of Mechanical Interface Mobilization Technique on Pain and Functional Status in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCRAHS-ISB/REC/MS-PT/017
Record Dates: First submitted 2024-04-29; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: CTS
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to the experimental group or control group. Participants were not notified which group was assigned to
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers who evaluated the participants were not informed of how the participants were grouped. Participants were informed that they would receive one of two different interventions without indicating which group should undergo mechanical interface mobilization technique or exercise therapy program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mechanical Interface Mobilisation Technique (Experimental): In the mechanical interface group, five techniques, including; wrist distraction (3 sets for 3 minutes), rhythmic and gentle stretching of the transverse carpal ligaments, release of palmar hand fascia, gliding of the finger flexor tendons (using oscillatory flexion-extension movement of metacarpophalangeal joint), and release of the upper forearm muscle and fascia will be applied. To release the upper forearm muscle as demonstrated for pronator teres muscle in, the therapist applied a firm pressure on the origin of the muscle by one thumb and concurrently moved the forearm into extension and supination (17).
  Interventions: Other: Mechanical Interface Mobilisation Technique
- Exercise Therapy (Active Comparator): Participants in this group will perform myofascial stretching of the carpal ligament, 3 days per week for four weeks along with isometric exercises at wrist joint as demonstrated by the physiotherapist.
  The participants will be instructed to perform gentle, pain-free isometrics of the wrist and hand musculature (25). Exercise would be performed with 5-10-second hold, with 10 repetitions (26).
  Interventions: Other: Exercise Therapy

INTERVENTIONS:
Other: Mechanical Interface Mobilisation Technique — In the mechanical interface group, five techniques, including; wrist distraction (3 sets for 3 minutes), rhythmic and gentle stretching of the transverse carpal ligaments, release of palmar hand fascia, gliding of the finger flexor tendons (using oscillatory flexion-extension movement of metacarpophalangeal joint), and release of the upper forearm muscle and fascia will be applied. To release the upper forearm muscle as demonstrated for pronator teres muscle in, the therapist applied a firm pressure on the origin of the muscle by one thumb and concurrently moved the forearm into extension and supination (17).
  Arms: Mechanical Interface Mobilisation Technique
Other: Exercise Therapy — Participants in this group will perform myofascial stretching of the carpal ligament, 3 days per week for four weeks along with isometric exercises at wrist joint as demonstrated by the physiotherapist.
  The participants will be instructed to perform gentle, pain-free isometrics of the wrist and hand musculature (25). Exercise would be performed with 5-10-second hold, with 10 repetitions (26).
  Arms: Exercise Therapy

SUMMARY:
The aim of this study is to find out the influence of mechanical interface mobilization technique which consists of 5 different steps, in management of carpal tunnel syndrome and how this technique effects pain and functional status in individuals who has carpal tunnel syndrome.

DETAILED DESCRIPTION:
The median nerve gets entrapped in the wrist, causing carpal tunnel syndrome (CTS), the most prevalent peripheral neuropathy in the upper limb. A number of clinical findings, such as sensory issues with the first three digits of the hand sensory distribution of the median nerve, a positive Phalen test, weakness and atrophy of the thenar muscle, and electrophysiological findings (prolonged motor and sensory distal latencies of the median nerve) are used to diagnose CTS . The most frequent occupational risk factors for CTS are repetitive wrist and finger motions or holding uncomfortable wrist positions for extended periods of time. Tenosynovitis of the finger flexors, a thicker transverse carpal ligament, a fracture or dislocation of the distal radius or lunate, rheumatoid arthritis, lipoma, diabetes, and hyperthyroidism are other non-occupational causes . A combination of techniques has been used in the studies of Seradge H. et al and Sucher Benjamin M. Et al which included mechanical interface and neuro-dynamics, but the isolated effects of each method is yet to be determined by further studies as their combined effects are more focused on in the current literature. And that leads to an unclear decision about, which group of manual therapy techniques has better effects on individuals suffering from CTS .

ELIGIBILITY:
Inclusion Criteria:

* Positive Phalen test and Tinel Test.
* Positive symptoms of CTS (Pain, numbness, or tingling in the first three and lateral half of the fourth finger.

Exclusion Criteria:

* No previous surgical treatments at the wrist joint, no fractures or open wounds at the wrist.
* Patients with thoracic outlet syndrome, and cervical radiculopathy.
* History of carpal tunnel release surgery.
* Steroid injection in the carpal tunnel.
* Pregnant females.
* Metabolic diseases such as diabetes, severe thyroid disorders and anemia.

Ages: 24 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 4 week (will be measured at the end of every week)]
  The VAS consists of a line, often 10 cm long, with verbal anchors at each end of the line, similar to a Numeric Rating Scale (i.e, no pain on the far left and severe pain on the far right). The patient places a mark at a point on the line corresponding to the patient's rating of pain intensity.
Symptom Severity Scale | 1st week(pre) and 4th week(post)]
  Symptom Severity Scale (SSS) (24) The SSS consists of 11 items related to six domains said to be critical for the evaluation of CTS.
  Each item is rated by the patient on a 1-5 (most severe) Likert scale, with higher ratings indicating more pain and disability.
Hand functional status scale | 1st week(pre) and 4th week(post)]
  Hand functional status scale (FSS) (24) The FSS consists of eight-items related to a variety of activities commonly performed by a diverse of patients. Each item is rated by the patient on a 1-5 (most severe) Likert scale, with higher ratings indicating more pain and disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ramsha Tariq, MsOMPT, Principal Investigator — Riphah International University
Locations (1):
- Dhqh Campus 2 Khushab, Khushāb, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chammas M, Boretto J, Burmann LM, Ramos RM, Dos Santos Neto FC, Silva JB. Carpal tunnel syndrome - Part I (anatomy, physiology, etiology and diagnosis). Rev Bras Ortop. 2014 Aug 20;49(5):429-36. doi: 10.1016/j.rboe.2014.08.001. eCollection 2014 Sep-Oct. PMID 26229841
- [Background] Michlovitz SL. Conservative interventions for carpal tunnel syndrome. J Orthop Sports Phys Ther. 2004 Oct;34(10):589-600. doi: 10.2519/jospt.2004.34.10.589. PMID 15552705
- [Background] Rota E, Morelli N. Entrapment neuropathies in diabetes mellitus. World J Diabetes. 2016 Sep 15;7(17):342-53. doi: 10.4239/wjd.v7.i17.342. PMID 27660694
- [Background] Naeser MA, Hahn KA, Lieberman BE, Branco KF. Carpal tunnel syndrome pain treated with low-level laser and microamperes transcutaneous electric nerve stimulation: A controlled study. Arch Phys Med Rehabil. 2002 Jul;83(7):978-88. doi: 10.1053/apmr.2002.33096. PMID 12098159
- [Background] Bland JD. Treatment of carpal tunnel syndrome. Muscle Nerve. 2007 Aug;36(2):167-71. doi: 10.1002/mus.20802. PMID 17534984
- [Background] Fernandez-de-Las Penas C, Ortega-Santiago R, de la Llave-Rincon AI, Martinez-Perez A, Fahandezh-Saddi Diaz H, Martinez-Martin J, Pareja JA, Cuadrado-Perez ML. Manual Physical Therapy Versus Surgery for Carpal Tunnel Syndrome: A Randomized Parallel-Group Trial. J Pain. 2015 Nov;16(11):1087-94. doi: 10.1016/j.jpain.2015.07.012. Epub 2015 Aug 15. PMID 26281946
- [Background] Kanaan N, Sawaya RA. Carpal tunnel syndrome: modern diagnostic and management techniques. Br J Gen Pract. 2001 Apr;51(465):311-4. PMID 11458486
- [Background] Zaralieva A, Georgiev GP, Karabinov V, Iliev A, Aleksiev A. Physical Therapy and Rehabilitation Approaches in Patients with Carpal Tunnel Syndrome. Cureus. 2020 Mar 3;12(3):e7171. doi: 10.7759/cureus.7171. PMID 32257712
- [Background] Huisstede BM, Hoogvliet P, Randsdorp MS, Glerum S, van Middelkoop M, Koes BW. Carpal tunnel syndrome. Part I: effectiveness of nonsurgical treatments--a systematic review. Arch Phys Med Rehabil. 2010 Jul;91(7):981-1004. doi: 10.1016/j.apmr.2010.03.022. PMID 20599038
- [Background] Jarvik JG, Comstock BA, Kliot M, Turner JA, Chan L, Heagerty PJ, Hollingworth W, Kerrigan CL, Deyo RA. Surgery versus non-surgical therapy for carpal tunnel syndrome: a randomised parallel-group trial. Lancet. 2009 Sep 26;374(9695):1074-81. doi: 10.1016/S0140-6736(09)61517-8. PMID 19782873
- [Background] Bialosky JE, Bishop MD, Price DD, Robinson ME, George SZ. The mechanisms of manual therapy in the treatment of musculoskeletal pain: a comprehensive model. Man Ther. 2009 Oct;14(5):531-8. doi: 10.1016/j.math.2008.09.001. Epub 2008 Nov 21. PMID 19027342
- [Background] Nijs J, Van Houdenhove B, Oostendorp RA. Recognition of central sensitization in patients with musculoskeletal pain: Application of pain neurophysiology in manual therapy practice. Man Ther. 2010 Apr;15(2):135-41. doi: 10.1016/j.math.2009.12.001. Epub 2009 Dec 24. PMID 20036180
- [Background] Lim YH, Chee DY, Girdler S, Lee HC. Median nerve mobilization techniques in the treatment of carpal tunnel syndrome: A systematic review. J Hand Ther. 2017 Oct-Dec;30(4):397-406. doi: 10.1016/j.jht.2017.06.019. Epub 2017 Jul 29. PMID 28764878
- [Background] Medina McKeon JM, Yancosek KE. Neural gliding techniques for the treatment of carpal tunnel syndrome: a systematic review. J Sport Rehabil. 2008 Aug;17(3):324-41. doi: 10.1123/jsr.17.3.324. PMID 18708684
- [Background] Burke J, Buchberger DJ, Carey-Loghmani MT, Dougherty PE, Greco DS, Dishman JD. A pilot study comparing two manual therapy interventions for carpal tunnel syndrome. J Manipulative Physiol Ther. 2007 Jan;30(1):50-61. doi: 10.1016/j.jmpt.2006.11.014. PMID 17224356
- [Background] Talebi GA, Saadat P, Javadian Y, Taghipour M. Manual therapy in the treatment of carpal tunnel syndrome in diabetic patients: A randomized clinical trial. Caspian J Intern Med. 2018 Summer;9(3):283-289. doi: 10.22088/cjim.9.3.283. PMID 30197774
- [Background] Talebi GA, Saadat P, Javadian Y, Taghipour M. Comparison of two manual therapy techniques in patients with carpal tunnel syndrome: A randomized clinical trial. Caspian J Intern Med. 2020;11(2):163-170. doi: 10.22088/cjim.11.2.163. PMID 32509244
- [Background] Akalin E, El O, Peker O, Senocak O, Tamci S, Gulbahar S, Cakmur R, Oncel S. Treatment of carpal tunnel syndrome with nerve and tendon gliding exercises. Am J Phys Med Rehabil. 2002 Feb;81(2):108-13. doi: 10.1097/00002060-200202000-00006. PMID 11807347
- [Background] Pinar L, Enhos A, Ada S, Gungor N. Can we use nerve gliding exercises in women with carpal tunnel syndrome? Adv Ther. 2005 Sep-Oct;22(5):467-75. doi: 10.1007/BF02849867. PMID 16418156
- [Background] Seradge H, Jia YC, Owens W. In vivo measurement of carpal tunnel pressure in the functioning hand. J Hand Surg Am. 1995 Sep;20(5):855-9. doi: 10.1016/S0363-5023(05)80443-5. PMID 8522756
- [Background] Sucher BM. Palpatory diagnosis and manipulative management of carpal tunnel syndrome. J Am Osteopath Assoc. 1994 Aug;94(8):647-63. PMID 7960973
- [Background] Ghasemi-Rad M, Nosair E, Vegh A, Mohammadi A, Akkad A, Lesha E, Mohammadi MH, Sayed D, Davarian A, Maleki-Miyandoab T, Hasan A. A handy review of carpal tunnel syndrome: From anatomy to diagnosis and treatment. World J Radiol. 2014 Jun 28;6(6):284-300. doi: 10.4329/wjr.v6.i6.284. PMID 24976931
- [Background] Oskouei AE, Talebi GA, Shakouri SK, Ghabili K. Effects of neuromobilization maneuver on clinical and electrophysiological measures of patients with carpal tunnel syndrome. J Phys Ther Sci. 2014 Jul;26(7):1017-22. doi: 10.1589/jpts.26.1017. Epub 2014 Jul 30. PMID 25140086
- [Background] Leite JC, Jerosch-Herold C, Song F. A systematic review of the psychometric properties of the Boston Carpal Tunnel Questionnaire. BMC Musculoskelet Disord. 2006 Oct 20;7:78. doi: 10.1186/1471-2474-7-78. PMID 17054773
- [Background] CAROLYN KISNER LACAJB. Therapeutic Exercises: Foundations and Techniques. 7th ed. Pine MADaJA, editor. Philadelphia PA, USA: F. A. Davis Company; 2018.
- [Background] McEvoy J, O'Sullivan K, Bron C. Therapeutic exercises for the shoulder region. Manual Therapy for Musculoskeletal Pain Syndromes: an evidence-and clinical-informed approach. 2015;373.